CLINICAL TRIAL: NCT06008574
Title: Cancer Anxiety Pilot Mindfulness Interdisciplinary Trial (CALM IT)
Brief Title: A Study Comparing Mindfulness Apps to Decrease Anxiety in People With Lung Cancer
Acronym: CALM IT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-114
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Anxiety; Mindfulness Apps; 23-114
MeSH Terms: conditions — Lung Neoplasms; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A prospective randomized pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCR (mindfulness-based cancer survivorship group) (AmDTx-PCSP) (Experimental): Patients randomized to the MBCR group will receive remote AmDTx-PCSP in the perioperative period (initiated at least 2 weeks before surgery). AmDTx-PCSP will be continued after surgery, for a minimum of 6 weeks total. AmDTx-PCSP is a step-by-step program including meditation training and other activities relevant for people living with cancer. The participants are asked to use AmDTx for about 20-30 minutes per day, at least 4 days per week, for 6 weeks. The participants are free to proceed at a faster pace and use AmDTx more than 20-30 per day if they choose. The first 3 modules of the program are required, and then the participant will be able to pick 3 additional modules based on topics that are most meaningful to them.
  Interventions: Other: AmDTx-PCSP; Other: Questionnaires
- CI (control) group (AmDTx-2048) (Active Comparator): Patients randomized to the CI group will use a game called "2048", a cognitive training app, which is used as an control condition to control for expectancy and daily engagement. The participants will use AmDTx-2048 to engage in cognitive training with a puzzle game. The participants are asked to use AmDTx for about 20-30 minutes per day, at least 4 days per week, for 6 weeks. The participants are free to proceed at a faster pace and use AmDTx more than 20-30 per day if you choose. In this puzzle game, the participants will slide numbered tiles around a grid, matching tiles of the same value to combine them into one new tile displaying the sum of the previous two numbers. The goal is to match tiles until the sum of 2048 is reached on a single tile. There is no time limit.
  Interventions: Other: AmDTx-2048; Other: Questionnaires

INTERVENTIONS:
Other: AmDTx-PCSP — Step-by-step program modules including meditation training and other activities relevant for people living with cancer
  Arms: MBCR (mindfulness-based cancer survivorship group) (AmDTx-PCSP)
Other: AmDTx-2048 — Cognitive training exercise called "2048".AmDTx-2048 is a modified version of a popular game called "2048. It is a fun and relaxing puzzle game". Within "2048", participants slide numbered tiles around a grid, matching tiles of the same value.
  Arms: CI (control) group (AmDTx-2048)
Other: Questionnaires — Distress Thermometer (DT)2, Demographic Information and medical history, Assessment for Contamination, Impact of Event Score (IES-R), Mindfulness Attention Awareness Scale (MAAS), PROMIS Short Form v1.0 - Anxiety - 8a, Depression - 4a, Fatigue 4a, Sleep Disturbance 4a, The Lung Cancer Stigma Inventory (LCSI)

SUMMARY:
The purpose of this study is to find out if it is practical to provide the program contained within the smartphone app AmDTx before and after lung cancer surgery. AmDTx is a platform that re-configures according to the specific needs of patients through physician prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lung cancer

  * Patients with suspected primary lung cancer per recent chest CT scan (with or without contrast) may be enrolled in the trial. These patients may be randomized and begin study intervention without a biopsy. If a patient undergoes a biopsy after consent and the results are negative or if the patient does not proceed with surgery, the patient will be removed from the study. The patient will continue to receive full access to the AmDTx app for 2-years.
  * Scheduled for surgery with at least 14 days lead time (to allow the participant to start the mindfulness practice [intervention group] 14 days preoperatively)
* Age ≥18 years of age at time of signing informed consent
* Access to a smartphone/tablet with data connection
* Willing to give time for mindfulness practice (Patients need to have the motivation to devote approximately 20 to 30 min daily, which is equal to 5 to 7 sessions a week over the course of a minimum of 6 weeks to do the mindfulness meditations and practices)
* Willing to be randomized to mindfulness MBCR or CI group and complete all assessments
* High distress level (Distress Thermometer score ≥4 at initial visit)
* Able to understand the study objectives and procedures, comply with the protocol, and sign an informed consent
* Able to read, speak, and understand English

Exclusion Criteria:

* Currently engaging in app-based mindfulness or meditation for one or more times per week
* As per self-report or as documented in the medical record, current untreated (e.g., no medication, no therapy) major psychotic disorder (schizotypal personality disorder, schizophreniform disorder, schizoaffective disorder). Patients diagnosed with a major psychiatric disorder will be reviewed by the study PI to determine eligibility before consent
* Individuals with impaired decision-making capacity
* Patients that need to undergo neoadjuvant therapy (chemotherapy±radiation)
* Patients undergoing active treatment of other non-lung cancers
* Patients with recurrent lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adherence Retention rate | up to 3 months
  Retention rates will be calculated separately as the proportion of enrolled participants who complete the 4-week and 3-month follow-up surveys. Adherence: The AmDTx app automatically collects adherence data, including date, time, length, and name of session to which participants listened, and transfers the data to the researchers on a weekly basis.

SECONDARY OUTCOMES:
Decrease in anxiety symptoms | up to 6 months
  These analyses apply to all continuous endpoints (PROMIS-Anxiety, IES, MAAS, PROMIS- Depression, PROMIS-Fatigue, PROMIS-Sleep Disturbance, LCSI)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Molena, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm